CLINICAL TRIAL: NCT03279705
Title: Division of Gastroenterology, Department of Internal Medicine, Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Chiayi, Taiwan
Brief Title: The efﬁcacy of the Integrated Water Jet Channel Colonoscopy in Water Exchange Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chih-wei Tseng (Other)
Responsible Party: Sponsor-Investigator, Chih-wei Tseng, Division of Gastroenterology, Department of Internal Medicine, Dalin Tzu Chi General Hospital
Organization: Dalin Tzu Chi General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DalinTCGH
Record Dates: First submitted 2017-08-24; First posted 2017-09-12 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Colonoscopy; Colon Disease
Keywords: water exchange; water jet channel colonoscopy; colonoscopy; cecal insertion time; adenoma detection rate
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Intervention Model Description: A total of 120 patients were allocated into one of two groups by computerized randomization. In group A (Two-channel group), clear water was infused through the water jet channel and dirty water was sucked form the accessy channel. In group B (One-channel group), water exchange was done by using the accessory channel for both infusing and suctioning of water.
Masking Description: These codes were contained in pre-arranged opaque envelopes, which were opened immediately before insertion of the colonoscope.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-channel group (Experimental): The colonoscopy was done with the new designed colonoscopy that integrated a separate water jet channel for infusing water. The dirty water was removed through other accessory channel.
  Interventions: Device: Water jet channel; Device: Accessory channel
- One-channel group (Active Comparator): The colonoscopy was done with the traditional colonoscopy. Water exchange was done by using the accessory channel for both infusing and suctioning of water.
  Interventions: Device: Accessory channel

INTERVENTIONS:
Device: Water jet channel — The separate water jet channel was used for infusing water.
  Arms: Two-channel group
Device: Accessory channel — The accessory channel was used for infusing and/or suctioning water

SUMMARY:
This prospective randomized controlled trial compared integrated water jet channel colonoscopy with traditional accessory channel colonoscopy in cecal insertion time among patients undergoing WE method colonoscopy.

DETAILED DESCRIPTION:
When the WE method colonoscopy were done with the accessory channel for both infusing and suctioning of water. The water had to be suctioned or infused alternatively and increaed the insertion time.

With the new designed endoscopy that integrated a separate water jet channel for infusing water, infusing and suctioning of water can be done at the same time. Besides, water jet pumping system could provide a powerful jet to help us open the collapse lumen and keep an appropriate distance between the mucosa and the lens, thus preventing loss of visualization. It will help the colonoscopist to find the way during insertion.

ELIGIBILITY:
Inclusion Criteria:

* Underwent fully sedative colonoscopy with WE method in the outpatient department

Exclusion Criteria:

* Age < 18 years old or > 80 years old
* Without standard colon preparation
* Allergy to meperidine or propofol
* With a history of partial colectomy
* Refusal to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
cecal insertion time | 2 hours
  Cecal insertion time was defined as the time from insertion into the rectum to the time when the colonoscope tip passed to a point proximal to the ileocecal valve so that the base of cecum was visible.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsi Hsieh, Study Director — Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tseng CW, Koo M, Hsieh YH. Cecal intubation time between the use of one-channel and two-channel water exchange colonoscopy: A randomized controlled trial. J Gastroenterol Hepatol. 2020 Sep;35(9):1562-1569. doi: 10.1111/jgh.15043. Epub 2020 Apr 6. PMID 32203986